CLINICAL TRIAL: NCT04265508
Title: Assessment of Hemostatic Profile in Patients With Mild to Advanced Liver Cirrhosis
Brief Title: Assessment of Hemostatic Profile in Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Elisabeth H. Adam, Division Chief of Critical Care, Goethe University
Other Study IDs: 195/17
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low MELD score: MELD score of 6 - 11
  Interventions: Other: Assessment of hemostatic profile
- High MELD score: MELD score of ≥ 17
  Interventions: Other: Assessment of hemostatic profile

INTERVENTIONS:
Other: Assessment of hemostatic profile — To assess the hemostatic profile, platelet function was analyzed by multiple electrode aggregometry (MEA) using Multiplate (ADP-, ASPI- and TRAP-test) and thrombelastometry using ROTEM (EXTEM, INTEM, FIBTEM)
  Other Names: Thrombelastometry; impedance aggregometry

SUMMARY:
Our study included both in- and outpatients suffering from liver cirrhosis attending the out- and inpatient care of the department of hepatology. Demographic and biochemical data as well as medical history including cause of liver cirrhosis, end stage kidney failure and medication with anticoagulants were recorded. To assess the hemostatic profile, platelet function was analyzed by multiple electrode aggregometry (MEA) using Multiplate (ADP-, ASPI- and TRAP-test) and thrombelastometry using ROTEM (EXTEM, INTEM, FIBTEM).

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* age of ≥ 18 years
* platelet count of at least 70 / nl

Exclusion Criteria:

* transfusion of platelet concentrate three weeks prior to inclusion
* pregnancy
* age < 18 years
* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attending the in- and outpatient care of the department of hepatology between 12/2017 and 05/2018 meeting the inclusion criteria were offered to participate in the present study. Inclusion criteria were liver cirrhosis and age of ≥ 18 years. Furthermore, a platelet count of at least 70 x103/µL was mandatory to ensure adequate measurement of MEA using the Multiplate analyzer. Patients were excluded when given a platelet concentrate three weeks prior to inclusion or in case of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Aggregation of platelets | Venous blood was collected via a cannula inserted into a cubital vein. Platelet function was measured by MEA using the Multiplate analyzer 15min after blood draw and after activation with commercially available standard reagents
  AUC of impedance aggregometry using multiple electrode aggregometry

SECONDARY OUTCOMES:
Viscoelastic measurements | Venous blood was collected via a cannula inserted into a cubital vein. Thrombelastometric assays were performed 15min after blood draw.
  Viscoelastic measurements of ROTEM assays (EXTEM, INTEM, FIBTEM)

CONTACTS AND LOCATIONS:
Locations (1):
- Universital Hospital Frankfurt / Main, Frankfurt am Main, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No